CLINICAL TRIAL: NCT06169306
Title: Do Throat Packs Used in Dental Treatments Under General anesthesıa of Patients With Special Health Care Needs Have an Effect on Ponv and Throat Pain?
Brief Title: Do Throat Pack Used in Dental Treatments Under General Anesthesia of Patients Have an Effect on PONV and Sore Throat?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sibel Tetiker, Lecturer, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUDHF-PABD
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Nausea and Vomiting; Sore-throat; Dental Caries
Keywords: PONV; sore throath; throath pack; special health care needs
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pharyngitis; Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Following endotracheal intubation, no throath pack will inserted into the hypopharynx.
- throath pack (Experimental): Following endotracheal intubation, throath pack will inserted into the hypopharynx.
  Interventions: Procedure: throat pack

INTERVENTIONS:
Procedure: throat pack — Following endotracheal intubation, one saline soaked, throat pack will inserted into the hypopharynx under direct vision. The packs will record in writting on the anaesthesia safety form.
  Arms: throath pack

SUMMARY:
The aim of this study is to investigate the effect of throat packs on PONV in dental treatments under general anesthesia in special health care needs.

DETAILED DESCRIPTION:
Throat packs are widely used to prevent aspiration of blood and other debris, especially in orofacial surgeries and dental treatments performed under general anesthesia. Aspiration of blood and other secretions into the stomach is one of the important causes of PONV. There is not much evidence that throat packs prevent nausea and vomiting after surgery. The most critical side effects of throat pack application are sore throat, difficulty swallowing, and being forgotten before extubation.

The incidence of cavities and other dental problems is higher in special health care needs due to reasons such as inadequate oral hygiene, malocclusion, high-carbohydrate diet, and lack of awareness about dental health. In this group of patients, dental treatments are primarily performed under general anesthesia. Since side effects are more difficult to identify by the patient, the procedures, technical applications and anaesthesia methods should be those with the least potential for side effects. Evidence is needed regarding the effect of throat packing on PONV. In this study, researchers planned to investigate the effects of using throat tampons during dental treatments under general anesthesia on PONV and sore throat in participants requiring special health care.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study with parental consent
* Being between the ages of 5-16
* Being grade 1 or 2 according to the ASA (American Society of Anesthesiologists) classification
* At least one primary or permanent and one restorative. Having undergone treatment (amalgam or composite restoration)

Exclusion Criteria:

* Having a tracheostomy
* Being evaluated as having difficult intubation
* Having an additional disease related to the oesophagus, stomach or intestines, having a percutaneous endoscopic gastrostomy,
* Having a history of PONV,
* Having morbid obesity,
* Having high airway pressure,
* Having a history of allergy to the drugs to be used,
* Needing an anaesthetic agent other than the anaesthesia method to be applied
* Having advanced mental retardation that prevents data collection

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
PONV | 1, 2 and 6 hours
  PONV scores were recorded at 1, 2 and 6 hours using the pictorial nausea scale "Baxter Retching Faces (BARF), which is scored between 0 and 10. A score of 0 on the BARF indicates the absence of PONV, while a score of 10 indicates the most severe PONV.

SECONDARY OUTCOMES:
sore throat | 1, 2 and 6 hours
  Sore throat scores were recorded at 1, 2 and 6 hours after endotracheal extubation, using the Visual Analog Scale (VAS) visual scale scored between 0 and 10. On the VAS, 0 indicates no pain, while 10 indicates the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Tetiker, Principal Investigator — Cukurova University Faculty of Dentistry, Pediatric Dentistry

REFERENCES:
- [Derived] Tetiker S, Akdogan HN, Alpay N, Dogan MC. Effect of Dental Throat Pack Used Under General Anesthesia in Children with Special Healthcare Needs on Postoperative Nausea, Vomiting, and Sore Throat: A Randomized Clinical Trial. J Clin Med. 2025 Jan 17;14(2):567. doi: 10.3390/jcm14020567. PMID 39860573